CLINICAL TRIAL: NCT00096382
Title: Treatment of Patients With Metastatic Melanoma Using a Transplant of Autologous Lymphocytes Reactive With Tumor Following a Myeloablative Lymphocyte Depleting Regimen of Chemotherapy, Total Body Irradiation and Reconstitution With CD34+ Cells
Brief Title: Cyclophosphamide, Fludarabine, and Total-Body Irradiation Followed By Cellular Adoptive Immunotherapy, Autologous Stem Cell Transplantation, and Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal investigator, National Institutes of Health Clinical Center (CC)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040288; 04-C-0288; NCI-7025; NCI-PRMC-P6273; CDR0000393480; NCT00092248 (obsolete NCT alias)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2; Filgrastim; Cyclophosphamide; fludarabine phosphate; Radiotherapy; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TBI 200cGy + TIL +HD IL-2, prior IL-2 (Other): Patients will receive 2Gy of total body irradiation (TBI) at a rate of 0.07 Gy/minute using a linear accelerator.
  Lymphocytes that that are isolated from the tumor, grown in the laboratory to high amounts and then infused into the patient.
  Interventions: Biological: aldesleukin; Biological: filgrastim; Biological: therapeutic tumor infiltrating lymphocytes; Drug: cyclophosphamide; Drug: fludarabine phosphate; Radiation: radiation therapy
- TBI 200cGy + TIL +HD IL-2, No prior IL-2 (Other): Patients will receive 2Gy of total body irradiation (TBI) at a rate of 0.07 Gy/minute using a linear accelerator.
  Lymphocytes that that are isolated from the tumor, grown in the laboratory to high amounts and then infused into the patient.
  Interventions: Biological: aldesleukin; Biological: filgrastim; Biological: therapeutic tumor infiltrating lymphocytes; Drug: cyclophosphamide; Drug: fludarabine phosphate; Radiation: radiation therapy

INTERVENTIONS:
Biological: aldesleukin — high dose: 720,000 IU/kg intravenously over 15 minutes every 8 hours for up to 5 days (maximum 5 doses) or low dose: 250,000 IU/kg subcutaneously daily for 5 days, after a two day rest, 125,000 IU/kg subcutaneously daily for 5 days for five weeks (2 days rest per week)
  Other Names: IL-2; Interleukin-2
Biological: filgrastim — 10 mcg/kg/day daily subcutaneously until neutrophil count >1x10^9/1.
  Other Names: GCSF
Biological: therapeutic tumor infiltrating lymphocytes — Lymphocytes that are isolated from the tumor, grown in the laboratory to high amounts and then infused into the patient.
Drug: cyclophosphamide — 60 mg/kg/day x 2 days intravenously over 1 hour
  Other Names: Cytoxan
Drug: fludarabine phosphate — 25 mg/m^2/day intravenous piggyback daily over 15-20 minutes for 5 days
  Other Names: Fludara
Radiation: radiation therapy — Patients will receive 2Gy of total body irradiation (TBI) at a rate of 0.07 Gy/minute using a linear accelerator.
  Other Names: total body irradiation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide and fludarabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Biological therapies, such as cellular adoptive immunotherapy, work in different ways to stimulate the immune system and stop tumor cells from growing. Autologous stem cell transplant may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy. Interleukin-2 may stimulate a person's lymphocytes to kill tumor cells. Combining chemotherapy, radiation therapy, and biological therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cyclophosphamide and fludarabine together with radiation therapy followed by cellular adoptive immunotherapy, autologous stem cell transplant, and interleukin-2 works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine complete clinical tumor regression in patients with metastatic melanoma treated with a myeloablative lymphoid-depleting preparative regimen comprising cyclophosphamide, fludarabine, and total body irradiation followed by autologous tumor-reactive tumor-infiltrating lymphocyte infusion, autologous CD34+ stem cell transplantation, and low-dose or high-dose interleukin-2.
* Evaluate the safety of this regimen in these patients.

Secondary

* Determine the survival of the infused lymphocytes by analyzing the sequence of the variable region of the T-cell receptor or flow cytometry in patients treated with this regimen.

OUTLINE:

* Autologous stem cell collection: Patients receive filgrastim (G-CSF) subcutaneously (SC) twice daily for 8 days. Beginning on day 5 of G-CSF, patients undergo apheresis daily for up to 3 days. Patients may receive 1 additional course of G-CSF and apheresis or use stem cells stored from a prior stem cell harvest in order to obtain an adequate number of cells.
* Lymphocyte-depleting myeloablative preparative regimen: Patients receive cyclophosphamide intravenous (IV) over 1 hour on days -5 and -6 and fludarabine IV over 15-30 minutes on days -6 to -2. Patients also undergo total body irradiation on day -1.
* Autologous lymphocyte infusion: Patients receive autologous tumor-reactive tumor-infiltrating lymphocytes IV over 20-30 minutes on day 0* followed by G-CSF SC once daily until blood counts recover.
* Autologous stem cell transplantation: Patients receive autologous CD34+ stem cells IV on day 2.
* Interleukin therapy: Patients are assigned to 1 of 2 cohorts, depending on whether they have received prior high-dose interleukin-2 (IL-2).

  * Cohort 1 (patients who received prior high-dose IL-2): Beginning on day 0*, patients receive high-dose IL-2 IV over 15 minutes 3 times daily for up to 5 days (maximum of 15 doses).
  * Cohort 3 (patients who have not received prior high-dose IL-2): Patients receive treatment as in cohort 1.

NOTE: *Day 0 is 1-4 days after the last dose of fludarabine.

Patients are evaluated at 4-6 weeks.

PROJECTED ACCRUAL: A total of 116 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma
* Measurable disease
* Resected or stable brain metastases are allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-1

Life expectancy

* At least 3 months

Hematopoietic

* See Immunologic
* Absolute neutrophil count > 1,000/mm^3 (without support of filgrastim [G-CSF])
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 8 g/dL (transfusion allowed)
* No coagulation disorders

Hepatic

* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 times upper limit of normal
* Bilirubin ≤ 2 mg/dL (< 3 mg/dL in patients with Gilbert's syndrome)
* No hepatitis B or C

Renal

* Creatinine ≤ 1.6 mg/dL

Cardiovascular

* Left ventricular ejection fraction (LVEF) ≥ 45% by cardiac stress test*
* No active major cardiovascular illness as evidenced by stress thallium or other comparable test
* No myocardial infarction
* No cardiac arrhythmias NOTE: *For patients ≥ 50 years of age receiving high-dose interleukin-2 (IL-2) OR patients with a history of electrocardiogram (EKG) abnormalities, symptoms of cardiac ischemia, or arrhythmias

Pulmonary

* Forced expiratory volume 1 (FEV_1) ≥ 60% of predicted by pulmonary function test in patients with prolonged history of cigarette smoking or symptoms of respiratory dysfunction*
* No active major respiratory illness
* No obstructive or restrictive pulmonary disease NOTE: *For patients receiving high-dose IL-2 only

Immunologic

* No active major immunologic illness
* No active systemic infections
* No primary or secondary immunodeficiency

  * Fully recovered immune competence after prior chemotherapy or radiotherapy as evidenced by both of the following:

    * Absolute neutrophil count > 1,000/mm^3
    * No opportunistic infections
* Human Immunodeficiency virus (HIV) negative
* Epstein-Barr virus positive

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 months after study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* At least 6 weeks since prior nitrosourea therapy
* No prior cyclophosphamide and fludarabine as part of a preparative regimen on National Cancer Institute (NCI) Surgery Branch adoptive cell therapy studies unless sufficient numbers of CD34+ stem cells (more than 2 x10^6/kg patient weight) have been obtained prior to the administration of chemotherapy

Endocrine therapy

* No concurrent systemic steroid therapy

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* Prior minor surgery within the past 3 weeks allowed if recovered

Other

* Recovered from all prior therapy
* At least 30 days since prior systemic therapy
* No other concurrent experimental agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Surgery Branch, Bethesda, Maryland

REFERENCES:
- [Derived] Yao X, Ahmadzadeh M, Lu YC, Liewehr DJ, Dudley ME, Liu F, Schrump DS, Steinberg SM, Rosenberg SA, Robbins PF. Levels of peripheral CD4(+)FoxP3(+) regulatory T cells are negatively associated with clinical response to adoptive immunotherapy of human cancer. Blood. 2012 Jun 14;119(24):5688-96. doi: 10.1182/blood-2011-10-386482. Epub 2012 May 3. PMID 22555974

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 34 participants who were enrolled, 8 patients were not assigned to treatment since their TIL did not grow. Of the 26 assigned to treatment, 1 patient was not actually treated therefore only 25 patients were evaluable.
Period: Overall Study
Arm/Group | TBI 200cGy + TIL +HD IL-2, Prior IL-2 | TBI 200cGy + TIL +HD IL-2, No Prior IL-2
Started | 23 | 3
Completed | 21 | 3
Not Completed | 2 | 0
Not completed — Not treated | 1 | 0
Not completed — Death during treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TBI 200cGy + TIL +HD IL-2, Prior IL-2 | TBI 200cGy + TIL +HD IL-2, No Prior IL-2 | Total
Number analyzed (Participants) | 23 | 3 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 3 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (9.6) | 48.3 (12.0) | 44.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 15 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 3 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 23 | 3 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Clinical Tumor Regression
Description: Tumor regression is defined as a complete response (CR) or partial response (PR) and was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is the disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Every 4-6 weeks for up to 1 year, and then every 6 months for up to 5 years.
Measure: Number; unit: Participants
Arm/Group | TBI 200cGy + TIL +HD IL-2, Prior IL-2 | TBI 200cGy + TIL +HD IL-2, No Prior IL-2
Number analyzed (Participants) | 23 | 3
Participants
  Complete Response | 1 | 1
  Partial Response | 9 | 2

2. Primary Outcome: Safety
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 4 years
Measure: Number; unit: Participants
Arm/Group | TBI 200cGy + TIL +HD IL-2, Prior IL-2 | TBI 200cGy + TIL +HD IL-2, No Prior IL-2
Number analyzed (Participants) | 23 | 3
Participants | 23 | 3

ADVERSE EVENTS:
Arm/Group | TBI 200cGy + TIL +HD IL-2, Prior IL-2 | TBI 200cGy + TIL +HD IL-2, No Prior IL-2
Serious Adverse Events (participants affected / at risk) | 3/22 | 1/3
Other Adverse Events (participants affected / at risk) | 22/22 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI 200cGy + TIL +HD IL-2, Prior IL-2 (N=22) | TBI 200cGy + TIL +HD IL-2, No Prior IL-2 (N=3)
Fatigue (General disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI 200cGy + TIL +HD IL-2, Prior IL-2 (N=22) | TBI 200cGy + TIL +HD IL-2, No Prior IL-2 (N=3)
Hemoglobin (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 17 (17) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 21 (21) | 3 (3)
Platelet (Blood and lymphatic system disorders) | 16 (16) | 3 (3)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Supraventricular & nodal arrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Vasovagal episode (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 8 (8) | 0 (0)
Rigors/Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (4) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (3) | 2 (2)
Insomnia (General disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Distention, bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 9 (9) | 3 (3) — fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever > =38.5 degrees C)
Infection (Infections and infestations) | 5 (5) | 0 (0)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 9 (9) | 1 (1)
ALT/SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
AST/SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (4) | 1 (2)
Creatinine (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Potassium, serum-high (hyperkalemia) increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Uric acid (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Apnea (Nervous system disorders) | 1 (1) | 0 (0)
Leak, Cerebrospinal fluid (CSF) (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Mood alteration (Nervous system disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 11 (11) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 22 (22) | 3 (3)
PTT (partial thromboplastin time) (Blood and lymphatic system disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No